CLINICAL TRIAL: NCT00185445
Title: A Phase II Study to Evaluate the Efficacy and Safety of Oral Fludarabine Phosphate in Combination With Mitoxantrone as First Line Treatment in Follicular NHL
Brief Title: Efficacy and Safety Study of Oral Fludarabine Phosphate in Combination With Mitoxantrone as First Line Treatment in Follicular NHL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 308580; 91381
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Non Hodgkin Lymphoma
Keywords: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Fludarabine Phosphate (Fludara)

INTERVENTIONS:
Drug: Fludarabine Phosphate (Fludara) — All patients will receive fludarabine phosphate orally for 3 consecutive days per cycle and mitoxantrone on day 1. Each patient will receive up to six treatment cycles. Treatment cycles will be given at 4 weeks intervals.
  Other Names: BAY86-4864

SUMMARY:
The purpose of the study is to demonstrate that oral fludarabine phosphate is comparable to i.v. formulation used in combination with mitoxantrone in terms of efficacy, safety and risk/benefit profile

DETAILED DESCRIPTION:
As of 29 May 2009, the clinical trial sponsor is Genzyme Corporation. NOTE: This study was originally posted by sponsor Schering AG, Germany, which was subsequently renamed to Bayer Schering Pharma AG, Germany.

ELIGIBILITY:
Inclusion Criteria:

* Indolent B-cell follicular non-Hodgkin's lymphoma (grade I-II according to REAL classification)
* Stage II to IV according to Ann Arbor staging system
* WHO performance status grade 0, 1 or 2 and life expectancy of greater than 6 months

Exclusion Criteria:

* Patients who have received any previous treatment for follicular NHL
* Patients with severe or life-threatening cardiac, pulmonary, neurological, psychiatric or metabolic disease
* Pregnant and lactating women
* Women of childbearing potential, and all men, not agreeing to take adequate contraceptive precautions during and for at least 6 months after cessation of therapy
* Laboratory screens positive for Hepatitis B, C or HIV infections
* Patients with autoimmune thrombocytopenia or hemolytic anemia with clinical evidence. NB. A positive Coombs test alone (with no clinical evidence of hemolysis) would not preclude entry in the study.
* Histological transformation to aggressive B-cell lymphoma
* Patients with prior malignancies except non melanoma skin tumors or stage 0 (in situ) cervical carcinoma
* Impairment of hepatic function unless disease related indicated by bilirubin, ASAT, ALAT or gamma-GT raised 2 times above the upper limit of the local laboratory range
* Impairment of renal function indicated by serum creatinine < 30 ml/min
* Patients who require systemic long-term therapy with glucocorticoids
* Participation at the same time in another study in which investigational drugs are used
* Patients unable to regularly attend outpatient clinic for treatment and assessments
* Any other co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent
* Patients with active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Complete response rate | Measurement of outcome 4 to 6 weeks after EOT

SECONDARY OUTCOMES:
Overall response rate, molecular response rate, toxicity profile, patients quality of life | Measurement of outcome 4 to 6 weeks after EOT

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (13):
- Italy (13):
  - Bologna, BO
  - Cesena, FC
  - Forlì, FC
  - Genova, GE
  - Roma, RM
  - Rimini, RN
  - Cagliari
  - Florence
  - Napoli
  - Ravenna
  - Roma
  - Siena
  - Udine